CLINICAL TRIAL: NCT02103816
Title: The Smartlipo Triplex 1440nm Wavelength Laser and the Sidelaze 800 Hand Piece for the Treatment of Facial Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-PRECIS-ACNE-BD
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Acne Scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SmartLipo Triplex laser system along with the SideLaze800 hand (Experimental)
  Interventions: Device: SmartLipo Triplex laser system along with the SideLaze800 hand piece

INTERVENTIONS:
Device: SmartLipo Triplex laser system along with the SideLaze800 hand piece

SUMMARY:
The purpose of this study to evaluate the SmartLipo Triplex laser system along with the SideLaze800 hand piece in the treatment of Acne Scars.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between 18 and 65 years old
* Has unwanted facial acne scars and wishes to undergo laser treatments.
* Is willing to consent to participate in the study.
* Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending follow up visits.

Exclusion Criteria:

* The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
* The subject is hypersensitive to light exposure OR takes photo sensitized medication.
* The subject has active or localized systemic infections.
* The subject has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to the heavy use of aspirin) {greater than 81 mg per day}).
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within the planned treatment area 3 months prior to entering this study.
* The subject has used Accutane within 6 months prior to enrollment.
* The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
* The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
* The subject has a history of keloids.
* The subject has evidence of compromised wound healing.
* The subject has a history of squamous cell carcinoma or melanoma.
* The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
* The subject has an allergy to lidocaine and epinephrine.
* The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- New Jersey Plastic Surgery, Montclair, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One additional patient was enrolled beyond the limitations specified by the original protocol. The protocol was amended (and approved by the IRB) part way through the study to allow for the enrollment of this additional subject.
Groups:
- SmartLipo Triplex Laser System Along With the SideLaze800 Hand: SmartLipo Triplex laser system along with the SideLaze800 hand piece
Period: Overall Study
Arm/Group | SmartLipo Triplex Laser System Along With the SideLaze800 Hand
Started | 21
Completed | 13
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | SmartLipo Triplex Laser System Along With the SideLaze800 Hand
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 8
  Race/Ethnicity: Asian | 2
  Race/Ethnicity: African American | 2
  Race/Ethnicity: Hispanic | 5
  Race/Ethnicity: Other | 4
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Score I | 0
    Fitzpatrick Skin Score II | 0
    Fitzpatrick Skin Score III | 11
    Fitzpatrick Skin Score IV | 7
    Fitzpatrick Skin Score V | 3
    Fitzpatrick Skin Score VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Facial Acne Improvement Using the Global Aesthetic Improvement Scale
Description: This assesses the level of improvement of acne scarring using the Global Aesthetic Improvement Scale. It is done through using photographic evaluation, comparing the baseline photograph to a photograph taken 3 months post the last treatment. The options for the acne scarring improvement are very much improved, much improved, improved, no change, or worse. The photographic evaluator decides this improvement based off of scar appearance differences amongst the photographs.
Time Frame: 3 months post treatment
Population: 1 subject completed the follow up over the phone, so there is no physician score for this subject. 2 subjects were a no-show for their appointment, but attended the other optional follow ups. The other 4 did not return to follow ups and could not be reached after numerous attempts to follow up.
Measure: Number; unit: percentage of participants
Arm/Group | SmartLipo Triplex Laser System Along With the SideLaze800 Hand
Number analyzed (Participants) | 14
percentage of participants
  Very Much Improved | 28.6
  Much Improved | 57.1
  Improved | 14.3

2. Secondary Outcome: Investigator Satisfaction Questionnaire
Description: The investigator chooses if they are extremely satisfied, satisfied, slightly satisfied, slightly dissatisfied, dissatisfied, or extremely dissatisfied with the results.
Time Frame: 3 months post treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SmartLipo Triplex Laser System Along With the SideLaze800 Hand
Number analyzed (Participants) | 14
Participants
  Extremely Satisfied | 6
  Satisfied | 5
  Slightly Satisfied | 3

3. Secondary Outcome: Subject Satisfaction Questionnaire
Description: The subject chooses if they are extremely satisfied, satisfied, slightly satisfied, slightly dissatisfied, dissatisfied, or extremely dissatisfied with the results.
Time Frame: 3 months post treatment
Population: 2 subjects were a no-show for their appointment, but attended the other optional follow ups. The other 4 did not return to follow ups and could not be reached after numerous attempts to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | SmartLipo Triplex Laser System Along With the SideLaze800 Hand
Number analyzed (Participants) | 15
Participants
  Extremely Satisfied | 6
  Satisfied | 6
  Slightly Satisfied | 2
  slightly dissatisfied | 1

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were captured and followed for the study duration, about 5 months.
Arm/Group | SmartLipo Triplex Laser System Along With the SideLaze800 Hand
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 16/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SmartLipo Triplex Laser System Along With the SideLaze800 Hand (N=21)
Pain (Nervous system disorders) | 2
Swelling (Skin and subcutaneous tissue disorders) | 15
Bruising (Skin and subcutaneous tissue disorders) | 3
Numbness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.